CLINICAL TRIAL: NCT00512824
Title: Calcium, Probiotics and Acute Diarrheal Disease Among Indonesian Children Aged 1-6 Years in Low Socio-economic Urban Area of East Jakarta
Brief Title: Calcium, Probiotics and Acute Diarrheal Disease Among Indonesian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other); SEAMEO-TROPMED RCCN University of Indonesia (Unknown)
Responsible Party: Ingeborg Bovee-Oudenhoven, Top Institute Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A011-CPDI
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Healthy; Diarrhea
Keywords: calcium; probiotics; diarrhea; children; Indonesia; Healthy children; acute diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: low calcium milk of 180 ml
- 2 (Active Comparator)
  Interventions: Dietary Supplement: regular milk of 180 ml
- 3 (Active Comparator)
  Interventions: Dietary Supplement: regular milk of 180 ml + probiotics
- 4 (Active Comparator)
  Interventions: Dietary Supplement: regular milk of 180 ml + probiotics

INTERVENTIONS:
Dietary Supplement: low calcium milk of 180 ml — twice daily for 24 weeks
  Arms: 1
Dietary Supplement: regular milk of 180 ml — twice daily for 24 weeks
  Arms: 2
Dietary Supplement: regular milk of 180 ml + probiotics — twice daily for 24 weeks
  Arms: 3
Dietary Supplement: regular milk of 180 ml + probiotics — twice daily for 24 weeks
  Arms: 4

SUMMARY:
This is a long term study on the efficacy of dietary calcium with or without probiotic strains in reducing the mean number of episodes and duration of diarrheal disease.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children aged 1-6 years, with emphasize on aged 2-5 years, living permanently in low socio-economic urban areas of East Jakarta for at least 6 months
* Parents are willing to sign the informed consent and give the supplements to the children for the period of 6 months
* Capable and willing to drink liquid milk with a straw (acceptance to be tested at screening by providing a sample drink and placebo straw to be consumed under supervision for 2 days)

Exclusion Criteria:

* Calcium intake exceeding 75% of the RDA for calcium (<375 mg/d) based on a Food Frequency Questionnaire
* Currently breastfed children
* Siblings of already included children that are living in the same household, except if it is a twin sibling
* Severely malnourished with or without oedema (Weight for height-WHZ Z-score of <-3.00 SD)
* Symptoms of chronic/congenital diseases and disabilities, suspected Tuberculosis by clinical examination, and /or history of allergic disease.
* Taking (any) antibiotics during 2 weeks prior to start of the study (children will be included after 3 weeks of last antibiotic intake
* Participation in another clinical trial at the same time or 2 months prior to the start of this study
* Both mothers and other caregivers present in the family are illiterate

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 494 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The mean number of episodes and duration of acute diarrheal disease | 24 weeks

SECONDARY OUTCOMES:
Incidence of acute diarrheal disease | 24 weeks
Severity of acute diarrheal disease | 24 weeks
Intestinal and systemic inflammation | 24 weeks
Intestinal colonization with pathogenic bacteria or viruses | 24 weeks
Nutritional status based on anthropometric measurement | 24 weeks
Iron and zinc status | 24 weeks
Incidence, mean episodes and duration of acute respiratory infections | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, MD, Principal Investigator — SEAMEO-TROPMED RCCN UI; Frans J. Kok, Prof, Study Chair — Division of Human Nutrition, Wageningen University (WUR); Ingeborg Bovee-Oudenhoven, PhD, Study Director — TIFN/ NIZO Food Research; Agus Firmansyah, Prof, MD, Study Chair — Faculty of Medicine University of Indonesia; Widjaja Lukito, MD, Study Director — SEAMEO-TROPMED RCCN UI
Locations (1):
- Seameo-Tropmed Rccn Ui, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Agustina R, Bovee-Oudenhoven IM, Lukito W, Fahmida U, van de Rest O, Zimmermann MB, Firmansyah A, Wulanti R, Albers R, van den Heuvel EG, Kok FJ. Probiotics Lactobacillus reuteri DSM 17938 and Lactobacillus casei CRL 431 modestly increase growth, but not iron and zinc status, among Indonesian children aged 1-6 years. J Nutr. 2013 Jul;143(7):1184-93. doi: 10.3945/jn.112.166397. Epub 2013 May 22. PMID 23700339
- [Derived] Agustina R, Kok FJ, van de Rest O, Fahmida U, Firmansyah A, Lukito W, Feskens EJ, van den Heuvel EG, Albers R, Bovee-Oudenhoven IM. Randomized trial of probiotics and calcium on diarrhea and respiratory tract infections in Indonesian children. Pediatrics. 2012 May;129(5):e1155-64. doi: 10.1542/peds.2011-1379. Epub 2012 Apr 9. PMID 22492764